CLINICAL TRIAL: NCT07002333
Title: Investigation of Respiratory Muscle Sarcopenia in Adults Diagnosed With Diabetes
Status: Not yet recruiting | Type: Observational
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Muhammed İhsan KODAK, assistant professor, Kirsehir Ahi Evran Universitesi
Other Study IDs: 2025-AEU-FTR-MK-01
Record Dates: First submitted 2025-04-25; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-04

CONDITIONS: Diabetes; Diabetes Mellitus; Sarcopenia; Atrophy
MeSH Terms: conditions — Diabetes Mellitus; Sarcopenia; Atrophy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with Diabetes: Individuals diagnosed with Type 2 Diabetes mellitus between the ages of 18-65

SUMMARY:
The aim of this study was to investigate respiratory muscle sarcopenia in individuals with diabet. The main question it aims to answer is:

What is the prevalence of respiratory muscle sarcopenia in patients with diabet? Participants body composition (bioelectrical impedance), hand grip strength (hand dynanometer), physical performance tests (5 repetition sit-and-stand test, 4-meter walk test, 6 minute walk test, Timed up-and-go test) and respiratory muscle strength were evaluated.

DETAILED DESCRIPTION:
The increase in the elderly population worldwide necessitates further research on age-related physiological changes and health problems related to these changes in geriatric individuals. One of these problems, sarcopenia, is a syndrome characterized by a decrease in muscle mass, muscle strength, and physical performance due to aging. Sarcopenia affects not only the extremity muscles but also the respiratory muscles, significantly reducing the individual's functional capacity and quality of life. Sarcopenia is a progressive and widespread loss of skeletal muscles, characterized by a decrease in muscle strength, muscle mass, and physical performance. Although it is usually seen in older individuals, it can also occur in people with certain diseases or who lead a sedentary lifestyle. The European Working Group on Sarcopenia in Older People (EWGSOP) has developed a guideline for the diagnosis of sarcopenia and determination of its severity. In line with this guideline, the EWGSOP considers sarcopenia in three basic stages: pre-sarcopenia, sarcopenia, and severe sarcopenia. Pre-sarcopenia is the stage in which muscle mass is low but muscle strength or physical performance is not yet affected. Sarcopenia is the stage in which low muscle mass is accompanied by decreased muscle strength or low physical performance. Severe sarcopenia is defined as the most advanced stage in which all these criteria are met. Respiratory muscle sarcopenia is defined as muscle fiber atrophy and weakness in the respiratory muscles. The Japanese Respiratory Sarcopenia Study Group defines this condition as whole-body sarcopenia with low respiratory muscle mass, decreased respiratory muscle strength, and/or respiratory dysfunction. Kera et al. (2019) evaluated respiratory muscle sarcopenia according to the peak expiratory flow rate value. However, whole-body sarcopenia and respiratory muscle strength are considered important parameters in the definition and diagnosis of respiratory muscle sarcopenia. It is reported that the rate of respiratory muscle sarcopenia is higher in the presence of sarcopenia. Sarcopenic respiratory failure is diagnosed in the presence of sarcopenia accompanied by functional disability, while individuals without functional disability but at risk for respiratory muscle sarcopenia are considered "at risk of sarcopenic respiratory failure". Sarcopenia is thought to be associated with insulin resistance and oxidative stress, leading to decreased muscle strength and muscle mass, as well as muscle atrophy. Respiratory muscles may also be affected in a similar way. Thus, weakening of respiratory muscles may lead to decreased respiratory function and decreased quality of life. In the current literature, studies examining the effects of aging on respiratory muscles are limited. Therefore, determining the potential effects of aging on respiratory muscles and evaluating respiratory muscle sarcopenia in this context may provide an important contribution to the development of new approaches and the literature.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65
* Diagnosed with Type 2 Diabetes mellitus
* Being clinically stable
* Ability to adapt to tests (visual, cognitive, cooperative)

Exclusion Criteria:

* Those with neurological and/or musculoskeletal problems that may affect the study
* Presence of severe joint contracture or painful ulcers that may affect muscle strength measurement and walking
* Presence of serious infection or sepsis
* Having a known additional rheumatological disease diagnosis
* Any stage of cancer
* Pregnant or breastfeeding women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sample size was calculated using G*Power Software (ver. 3.1.3.2). A similar study in the literature was taken as a basis. The measurement values of the similar study were used to calculate the effect size (Effect size (d) = 0.12). Accordingly, the sample size of the study was found to be 84 participants with a 5% margin of error and 80% power.
Sampling Method: Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Respiratory Muscle Sarcopenia Assessment | Baseline
  The diagnosis of respiratory muscle sarcopenia will also be made by combining the results of secondary measurements.
  Participants included in the study:
  Hand grip strength <27 kg for men and <16 kg for women, Bioelectrical Impedance Analysis (Skeletal muscle mass (SMM) <20 kg for men and <15 kg for women) the participant is diagnosed with sarcopenia. They will also be diagnosed with a frailty phenotype based on the results of the Timed Stand and Walk Test, the 4 meter walk test and the 5 Repetition Sit and Stand Test.
  Patients diagnosed with sarcopenia will be diagnosed with respiratory muscle sarcopenia if respiratory muscle weakness is also detected.

SECONDARY OUTCOMES:
Body composition | baseline
  Body mass and body composition will be measured using bioelectrical impedance method. The variables to be assessed are body mass index (BMI = body mass (kg)/height2 (m)2 ), fat mass (pFM) expressed as a percentage of body mass, fat-free mass (FFM) expressed in kilograms, and appendicular skeletal muscle mass (ASMM) and skeletal muscle mass (SMM) expressed in kilograms. Data will be collected with a bioelectrical impedance device and recorded on pre-prepared forms. The measurement will be made with a Tanita brand device. All measurement results will be obtained from the measurement report given by the device.
Grip Force Measurement | baseline
  The hand muscle grip strength of the individuals will be measured with a hand dynamometer. During the measurement, the position recommended by the American Association of Hand Therapists (ASHT); the participant will be in an upright sitting position and no arm support will be allowed on the sitting surface. The elbow and knee angle will be set to 90°. The wrist will be held without deviation. The measurement will be performed 3 times with an interval of 10 seconds and the highest value will be used in the study.
5 Repetition Sit and Stand Test | baseline
  An armless chair with a straight back support and a rigid seat at a height of 48 cm from the floor will be fixed to the wall. Participants will be asked to sit on the chair and come forward in the chair until their feet are flat on the floor. Participants will be asked to do a "stand and sit" movement once with their arms crossed across their chest. The test will be terminated for those who cannot complete the task or need assistance. Those who successfully complete the first task will be asked to perform five consecutive stand and sit as fast as possible. The timing is started with the command start and stopped at the end of the fifth posture. Our participants test scores will be recorded in seconds using a stopwatch.
4 Meter Walking Speed Test (4MWT) | baseline
  4MWT is a measure of walking speed, a vital sign of mobility and functionality. In older adults, walking speed is a clinical indicator of conditions such as frailty and sarcopenia. Participants were instructed to start walking at their normal speed 2 m behind the "start point" and continue until they passed the "end point". Using a stopwatch, the time taken for each participant to walk the 4 m distance between the "start" and "end" point will be measured. This will be used to calculate walking speed (distance/time).
Timed Up and Go Test (TUG) | baseline
  This functional test measures the time it takes for an individual to stand up from a standard chair, walk 3 m at normal speed, turn around, walk back to the starting point and sit down. Using a stopwatch, participants test scores are recorded in seconds.
Respiratory muscle strength | baseline
  Intraoral pressure will be measured with a measuring device. They are easily applicable and simple measurements. Maximal voluntary inspiratory and expiratory pressures (MIP and MEP) are the most commonly used noninvasive methods to measure respiratory muscle strength. It is based on Müller (maximal inspiration) and Valsalva (maximal expiration).
6 Minute Walk Test (6MWT): | baseline
  The 6-minute walk test is used as a simple measure of aerobic exercise and functional capacity. During this test, a 30-meter track with a hard surface is walked at a normal pace for six minutes. This track is marked every 3 meters and a cone is placed at the end of this 30-meter track and the same track is returned around it. During the test, participants must walk at a speed appropriate to their condition and are allowed to stop or slow down if they wish and continue walking as soon as possible. Initial oxygen saturation, heart rate and blood pressure are measured. In addition, the Borg scale rating is used for shortness of breath and fatigue.
Age | Baseline
  Age will be questioned and data will be recorded on pre-prepared forms.
Height | Baseline
  Height(meter) will be questioned and data will be recorded on pre-prepared forms.
Gender | Baseline
  Gender will be questioned and data will be recorded on pre-prepared forms.
Educational status | Baseline
  Educational status will be questioned and data will be recorded on pre-prepared forms.
Medication use | Baseline
  Medication use will be questioned and data will be recorded on pre-prepared forms.

IPD SHARING:
Plan to Share IPD: No